CLINICAL TRIAL: NCT02447055
Title: Allogeneic Stem Cell Transplantation for Patients With Multiple Myeloma: a Pilot Feasibility Study Using a Novel Protocol
Brief Title: Allogeneic Stem Cell Transplantation for Patients With Multiple Myeloma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201508102
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma; Myeloma-Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab; Melphalan; fludarabine; fludarabine phosphate; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Flu/Mel/PT-Cy & Tac/MMF for certain cases) (Experimental): * Fludarabine 30 mg/m^2 intravenously (IV) on Days -5, -4, -3, and -2
  * Melphalan 140 mg/m^2 IV on Day -2
  * Tocilizumab 8 mg/m^2 (capped at 800 mg) IV on Day -1
  * Stem cell infusion on Day 0
  * Cyclophosphamide 50 mg/kg IV on Days +3 and +4
  * Tacrolimus 1 mg/day IV on Day +5 (for unrelated & haploidentical cases)
  * Mycophenolate mofetil 15 mg/kg orally three times per day on Day +5 (for unrelated & haploidentical cases)
  * Filgrastim 10 ug/kg/day subcutaneously until neutrophil recovery starting on Day +5
  Interventions: Biological: Tocilizumab; Drug: Melphalan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Filgrastim

INTERVENTIONS:
Biological: Tocilizumab
  Other Names: Actemra®
Drug: Melphalan
  Other Names: Alkeran®; Phenylalanine mustard
Drug: Fludarabine
  Other Names: Fludara®; 2-Fluoro-ara-A Monophosphate; 2-Fluoro-ara AMP; FAMP
Drug: Cyclophosphamide
  Other Names: Cytoxan®; CPM; CTX; CYT
Drug: Tacrolimus
  Other Names: Prograf®; FK-506
Drug: Mycophenolate mofetil
  Other Names: CellCept®; Myfortic®
Drug: Filgrastim
  Other Names: Granix®; Neupogen®; Granulocyte Colony-Stimulating Factor; G-CSF; Recombinant Methionyl Human G-CSF

SUMMARY:
The purpose of this study is to develop a novel platform for allo-SCT in multiple myeloma (MM) with the idea of maximizing anti-myeloma effect with conditioning and minimizing GvHD (graft versus host disease). Specifically, the investigators will use the Flu/Mel (fludarabine and melphalan) regimen. For GvHD prophylaxis, the investigators use the Hopkins PT-Cy (post-transplant cyclophosphamide) platform with the novelty of adding tocilizumab as both an anti-myeloma therapy and as a method to reduce GvHD. IL-6 has an important role in promoting the growth of myeloma cells and progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of myeloma.
* Between 18 and 70 years of age (inclusive).
* Karnofsky performance status ≥ 50% or ECOG performance score of ≤ 2 -Completion of last anti-myeloma therapy (if any) must occur at least 14 days before conditioning.
* Must have an HLA-matched sibling, HLA-matched unrelated donor, or a related haploidentical donor:
* Available HLA-matched sibling or unrelated donor must meet the following criteria:

  * At least 18 years of age
  * HLA donor/recipient match based on at least low-resolution typing per institutional standards (syngeneic donors [identical twins] are excluded)
  * In the investigator's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting stem cells
  * No active hepatitis
  * Negative for HTLV and HIV
  * Not pregnant

OR

* Available haploidentical donor must meet the following criteria:

  * Blood-related family member (sibling (full or half), offspring, parent, cousin, niece or nephew, aunt or uncle, or grandparent)
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by at least low-resolution typing per institutional standards
  * In the investigator's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting stem cells
  * No active hepatitis
  * Negative for HTLV and HIV
  * Not pregnant
* Normal bone marrow and organ function as defined below within 14 days prior to first study drug dose (conditioning regimen):

  * Total bilirubin ≤ 2.5 mg/dl
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
  * Creatinine ≤ 2.0 x ULN OR estimated creatinine clearance ≥ 30 mL/min/1.73 m2 by Cockcroft-Gault Formula (See Appendix C)
  * Oxygen saturation ≥ 90% on room air
  * LVEF ≥ 40%
  * FEV1 and FVC ≥ 40% predicted, DLCOc ≥ 40% predicted
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry through Day +100 visit. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Receiving renal replacement therapy, hemodialysis, or peritoneal dialysis.
* Presence of another concurrent malignancy requiring treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan, cyclophosphamide, or other agents used in the study.
* Presence of an uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding.
* Previous treatment with tocilizumab (TCZ).
* Immunization with a live/attenuated vaccine within 28 days prior to conditioning.
* Any history of recent serious bacterial, viral, fungal, or other opportunistic infections, precluding a stem cell transplant according to the treating physician.
* Serologic evidence of HIV
* Active infection with Hepatitis A, B, or C. Active infection is defined as serologic positivity and elevated liver function tests.
* History of tuberculosis
* Active infection with EBV as defined as EBV viral load ≥ 10,000 copies per mL of whole blood; EBV viral load testing is only required if the patient has clinical signs or symptoms suggestive of active EBV infection
* Active infection with CMV as defined as CMV viral load ≥ 10,000 copies per mL of whole blood; CMV viral load testing is only required if the patient has clinical signs or symptoms suggestive of active CMV infection
* History of complicated diverticulitis, including fistulae, abscess formation or gastrointestinal (GI) perforation.
* Pre-existing CNS demyelination or seizure disorders
* Major surgery within preceding 8 weeks
* Body weight >150kg
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of regimen as measured by grade and frequency of adverse events | Day +100
  Adverse events will be graded using NCI CTCAE v4.0 and summarized by grade and frequency

SECONDARY OUTCOMES:
Cumulative incidence and severity of acute GvHD | 6 months
Cumulative incidence and severity of chronic GvHD | 1 year
Non-relapse mortality (NRM) | 1 year
  -NRM is defined as death occurring in a patient from causes other than disease relapse or progression
Non-relapse mortality (NRM) | Day +100
  -NRM is defined as death occurring in a patient from causes other than disease relapse or progression
Progression-free survival (PFS) | 1 year
  -PFS is defined as the duration from transplant to time of first progression, death, relapse after CR, or the date the patient was last known to be in remission.
Overall survival (OS) | 1 year
  -OS is defined as the duration from the time of transplant to death or last follow-up.
Time to neutrophil engraftment | Day +30
  * Neutrophil engraftment is defined as ANC > 0.5 × 10^9/L × 3 consecutive daily assessments. The first of 3 consecutive days for which ANC > 0.5 × 10^9/L will be recorded as the date of neutrophil engraftment. Time to neutrophil engraftment will be calculated as the time from the date of the ASCT to the date of neutrophil engraftment.
  * Non-engraftment is defined as failure to reach an ANC > 0.5 × 10^9/L × 3 consecutive daily assessments by Day +30.
Time to platelet engraftment | Day +100
  * Platelet engraftment is defined as an untransfused platelet measurement > 20,000/ x10^9/L × 3 consecutive daily assessments. The first of 3 consecutive days for which the untransfused platelet measurement is > 20,000 x 10^9/L will be recorded as the date of platelet engraftment. Time to platelet engraftment will be calculated as the time from receiving the date of ASCT to the date of platelet engraftment. Untransfused is defined as no transfusions within 7 days.
  * Non-engraftment is defined as failure to reach platelets > 20,000 × 10^9/L × 3 consecutive assessments by Day +100.
Non-relapse mortality (NRM) | Day +180
  -NRM is defined as death occurring in a patient from causes other than disease relapse or progression

CONTACTS AND LOCATIONS:
Overall Officials: John F DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu